CLINICAL TRIAL: NCT01782326
Title: A 52-week Treatment, Multi-center, Randomized, Double-blind, Double Dummy, Parallel-group, Active Controlled Study to Compare the Effect of QVA149 (Indacaterol Maleate / Glycopyrronium Bromide) With Salmeterol/Fluticasone on the Rate of Exacerbations in Subjects With Moderate to Very Severe COPD. (FLAME).
Brief Title: QVA vs. Salmeterol/Fluticasone, 52-week Exacerbation Study, FLAME (EFfect of Indacaterol Glycopyronium Vs Fluticasone Salmeterol on COPD Exacerbations)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQVA149A2318
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, QVA149, FLAME( EFfect of Indacaterol Glycopyronium Vs Fluticasone salmeterol on COPD Exacerbations)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 (Experimental): QVA149 (110/50 μg) once daily
  Interventions: Drug: QVA149
- Long acting B2 agonist (LABA) and inhaled corticosteroid (ICS) (Active Comparator): Salmeterol/fluticasone (50/500μg) b.i.d
  Interventions: Drug: Long acting B2 agonist (LABA) and inhaled corticosteroid (ICS)

INTERVENTIONS:
Drug: QVA149 — QVA149 will be supplied in a capsule form in blister packs for use in the Novartis Concept 1 SDDPI.
  Arms: QVA149
Drug: Long acting B2 agonist (LABA) and inhaled corticosteroid (ICS) — Salmeterol/fluticasone dry inhalation powder delivered via the Accuhaler device.
  Arms: Long acting B2 agonist (LABA) and inhaled corticosteroid (ICS)

SUMMARY:
This study will assess the efficacy, safety and tolerability of QVA149 in patients with moderate to very severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Male or female adults aged ≥40 years
* Patients with stable Chronic Obstructive Pulmonary Disease ( COPD) according to the current GOLD strategy (GOLD 2011)
* Current or ex-smokers who have a smoking history of at least 10 pack years. (Ten pack-years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years)
* Patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) ≥25 and < 60% of the predicted normal value, and post-bronchodilator FEV1/FVC (Forced Vital Capacity) < 0.70 at day -28. (Post refers to 1 hour after sequential inhalation of 84 µg (or equivalent dose) of ipratropium bromide and 400 µg of salbutamol)
* A documented history of at least 1 COPD exacerbation in the previous 12 months that required treatment with systemic glucocorticosteroids and/or antibiotics
* Patients taking stable COPD medication (at least 60 days) prior to day 28
* Patients with an mMRC grade of at least 2 at day 28

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG (human Chorionic Gonadotropin) laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Patients with Type I or uncontrolled Type II diabetes
* Patients with a history of long QT syndrome or whose QTc measured at day 28 (Fridericia method) is prolonged (>450 ms for males and females) and confirmed by a central assessor. These patients should not be re-screened
* Patients who have a clinically significant ECG abnormality prior to randomization. (These patients should not be re-screened)
* Patients who have a clinically significant laboratory abnormality at screening
* Patients who have clinically significant renal, cardiovascular (such as but not limited to unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, myocardial infarction), arrhythmia (see below for patients with atrial fibrillation), neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological abnormalities which could interfere with the assessment of the efficacy and safety of the study treatment
* Patients with paroxysmal (e.g. intermittent) atrial fibrillation are excluded
* Patients with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., selective beta blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) for at least 6 months may be considered for inclusion. In such patients, atrial fibrillation must be present at both pre-randomization visits, with a resting ventricular rate < 100/min. At screening the atrial fibrillation must be confirmed by central reading
* Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof: anticholinergic agents, long and short acting beta-2 agonists, sympathomimetic amines, lactose or any of the other excipients of trial medication
* Patients with a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment or urinary retention. Benign Prostatic Hyperplasia (BPH) patients who are stable on treatment can be considered
* Patients who have not achieved an acceptable spirometry results at screening in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria for acceptability (one retest may be performed for patients that don't meet the acceptability criteria)
* Patients who have had a COPD exacerbation that required treatment with antibiotics and/or systemic corticosteroids and/or hospitalization in the 6 weeks prior to screening
* Patients who develop a COPD exacerbation of any severity (mild/moderate/severe) between screening and treatment will not be eligible but will be permitted to be re-screened after a minimum of 6 weeks after the resolution of the COPD exacerbation
* Patients who have had a respiratory tract infection within 4 weeks prior to screening
* Patients who develop a respiratory tract infection between screening and prior to treatment will not be eligible, but will be permitted to be re-screened 4 weeks after the resolution of the respiratory tract infection
* Patients requiring long term oxygen therapy prescribed for >12 hours per day
* Patients with any history of asthma
* Patients with an onset of respiratory symptoms, including a COPD diagnosis prior to age 40 years
* Patients with a blood eosinophil count > 600/mm3 at screening
* Patients with allergic rhinitis who use a H1 antagonist or intra-nasal corticosteroids intermittently (treatment with a stable dose or regimen is permitted)
* Patients with concomitant pulmonary disease (e.g. lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension)
* Patients with clinically significant bronchiectasis
* Patients with a diagnosis of α-1 anti-trypsin deficiency
* Patients with active pulmonary tuberculosis, unless confirmed by imaging to be no longer active
* Patients with pulmonary lobectomy or lung volume reduction surgery or lung transplantation
* Patients participating in or planning to participate in the active phase of a supervised pulmonary rehabilitation program during the study. (Maintenance program is permitted.)
* Patients receiving any medications in the classes listed in the protocol
* Patients receiving any COPD related medications in the classes specified in the protocol must undergo the required washout period prior to screening and follow the adjustment to treatment program
* Use of other investigational drugs/devices (approved or unapproved) at the time of enrollment, or within 30 days or 5 half-lives of screening, whichever is longer
* Patients unable to use an electronic patient diary and EXACT pro diary
* Patients unable to use a dry powder inhaler device, Metered Dose Inhaler (MDI) or a pressurized MDI (rescue medication) or comply with the study regimen.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3362 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (427):
- Argentina (12):
  - Novartis Investigative Site, Ciudad de Buenos Aires, Argentina
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Austria (10):
  - Novartis Investigative Site, Feldbach, Austria
  - Novartis Investigative Site, Feldkirch, Austria
  - Novartis Investigative Site, Graz, Austria
  - Novartis Investigative Site, Grieskirchen, Austria
  - Novartis Investigative Site, Linz, Austria
  - Novartis Investigative Site, Thalheim bei Wels, Austria
  - Novartis Investigative Site, Wels, Austria
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (15):
  - Novartis Investigative Site, Gosselies, BEL
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Luxembourg, Luxembourg
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Gilly
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Ostend
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Wavre
- Bulgaria (9):
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Troyan Municipality
- Canada (11):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Downsview, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Charles-Borromée, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Chile (3):
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Quillota
  - Novartis Investigative Site, Santiago
- China (18):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (4):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Medellín
- Croatia (3):
  - Novartis Investigative Site, Zagreb, Croatia
  - Novartis Investigative Site, Karlovac
  - Novartis Investigative Site, Zagreb
- Czechia (15):
  - Novartis Investigative Site, Cvikov, Czech Republic
  - Novartis Investigative Site, Český Krumlov, Czech Republic
  - Novartis Investigative Site, Jindrichuv Hradec III, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Mělník, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Ostrava - Hrabuvka, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Praha 6 - Repy, Czech Republic
  - Novartis Investigative Site, Strakonice, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Žatec, Czech Republic
  - Novartis Investigative Site, Benešov
  - Novartis Investigative Site, Olomouc
- Denmark (9):
  - Novartis Investigative Site, Aalborg, Denmark
  - Novartis Investigative Site, Hellerup, Denmark
  - Novartis Investigative Site, Hvidovre, Denmark
  - Novartis Investigative Site, Roskilde, Denmark
  - Novartis Investigative Site, Silkeborg, Denmark
  - Novartis Investigative Site, Sønderborg, Denmark
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Næstved
- Estonia (2):
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Tallinn
- Finland (6):
  - Novartis Investigative Site, Turku, Finland
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, HUS
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Pori
- France (11):
  - Novartis Investigative Site, Beuvry, France
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Briis-sous-Forges
  - Novartis Investigative Site, Cournonterral
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Saint-Génis-des-Fontaines
- Germany (54):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Dresden, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Marburg, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Geesthacht, Schleswig-Holstein
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Delitzsch
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freudenberg
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hannover Münden
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Oranienburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien A. Chiemsee
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Schwabach
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Teuchern
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Warendorf
  - Novartis Investigative Site, Weinheim
  - Novartis Investigative Site, Wissen
  - Novartis Investigative Site, Witten
- Greece (9):
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Serres, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Rethymno, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion Crete
  - Novartis Investigative Site, Thessaloniki
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, Departamento de Guatemala
  - Novartis Investigative Site, Ciudad, Gautemala
- Hong Kong (2):
  - Novartis Investigative Site, Kowloon, Hong Kong
  - Novartis Investigative Site, New Territories, Hong Kong
- Hungary (4):
  - Novartis Investigative Site, Komárom, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Törökbálint
- Novartis Investigative Site, Reykjavik, Iceland
- India (12):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Vijayawada, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Bangalore
- Italy (18):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cassano delle Murge, BA
  - Novartis Investigative Site, Crema, CR
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavullo nel Frignano, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Cittadella, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Cuasso al Monte, VA
  - Novartis Investigative Site, Tradate, VA
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Napoli
- Japan (26):
  - Novartis Investigative Site, Komaki, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Kōshi, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Matsusaka, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Iwata, Shizuoka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
- Latvia (3):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (7):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Vilnius, LT
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Mexico (6):
  - Novartis Investigative Site, Aguascalientes, Aguascalientes
  - Novartis Investigative Site, Guadalajara Jalisco, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Puebla City, Puebla
  - Novartis Investigative Site, Mexico City
- Netherlands (9):
  - Novartis Investigative Site, Almelo, Netherlands
  - Novartis Investigative Site, Enschede, Netherlands
  - Novartis Investigative Site, Harderwijk, Netherlands
  - Novartis Investigative Site, Zutphen, Netherlands
  - Novartis Investigative Site, Assen
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Geldrop
  - Novartis Investigative Site, Groningen
- Norway (8):
  - Novartis Investigative Site, Follebu
  - Novartis Investigative Site, Hønefoss
  - Novartis Investigative Site, Kløfta
  - Novartis Investigative Site, Kongsvinger
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Svelvik
  - Novartis Investigative Site, Trondheim
- Philippines (3):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Bulacan, Philippines
  - Novartis Investigative Site, Quezon City
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Piła
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Wroclaw
- Portugal (11):
  - Novartis Investigative Site, Lisbon, Lisbon District
  - Novartis Investigative Site, Almada, Portugal
  - Novartis Investigative Site, Barcelos, Portugal
  - Novartis Investigative Site, Braga, Portugal
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Lisbon, Portugal
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Torres Vedras, Portugal
  - Novartis Investigative Site, Vila Franca de Xira, Portugal
  - Novartis Investigative Site, Vila Nova de Gaia, Portugal
  - Novartis Investigative Site, Viseu, Portugal
- Romania (15):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Brasov, Romania
  - Novartis Investigative Site, Bucharest, Romania
  - Novartis Investigative Site, Deva, Romania
  - Novartis Investigative Site, Iași, Romania
  - Novartis Investigative Site, Oradea, Romania
  - Novartis Investigative Site, Târgu Mureş, Romania
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Deva
- Russia (10):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yaroslavl
- Serbia (3):
  - Novartis Investigative Site, Belgrade, Serbia
  - Novartis Investigative Site, Knez-Selo
  - Novartis Investigative Site, Kragujevac
- Slovakia (16):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Partizánske, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Lučenec, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Považská Bystrica, Slovakia
  - Novartis Investigative Site, Námestovo, Slovensko
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Spisská Nová Ves
- South Africa (7):
  - Novartis Investigative Site, Berea, Durban
  - Novartis Investigative Site, Sandton, Gauteng
  - Novartis Investigative Site, Pretoria, South Africa
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Gatesville
  - Novartis Investigative Site, Port Elizabeth
  - Novartis Investigative Site, Pretoria
- South Korea (6):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Jeonju, Jeollabuk-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (19):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Torrelavega, Cantabria
  - Novartis Investigative Site, Burgos, Castille and León
  - Novartis Investigative Site, Ponferrada, Castille and León
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Salt, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Cartagena, Murcia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
- Sweden (6):
  - Novartis Investigative Site, Borås
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Trollhättan
  - Novartis Investigative Site, Uddevalla
- Taiwan (7):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei County, Taiwan
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Chiayi County
  - Novartis Investigative Site, Niaosong Township
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (4):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kinikli / Denizli
  - Novartis Investigative Site, Manisa
  - Novartis Investigative Site, Mersin
- United Kingdom (19):
  - Novartis Investigative Site, Huntingdon, Cambridgeshire
  - Novartis Investigative Site, Stockton, Cleveland
  - Novartis Investigative Site, Midsomer Norton, Radstock
  - Novartis Investigative Site, Axbridge, Somerset
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, South Shields, Tyne and Wear
  - Novartis Investigative Site, Cambridge, United KIngdom
  - Novartis Investigative Site, Crawley, West Sussex
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Chester
  - Novartis Investigative Site, Darlington
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Tyne & Wear
  - Novartis Investigative Site, Wiltshire

REFERENCES:
- [Derived] Mathioudakis AG, Bate S, Chatzimavridou-Grigoriadou V, Sivapalan P, Jensen JS, Bakerly ND, Vestbo J, Singh D. Disproportionate increase in COPD exacerbation risk for 3 months after discontinuing LAMA or ICS: insights from the FLAME trial. Thorax. 2025 Dec 15:thorax-2025-223282. doi: 10.1136/thorax-2025-223282. Online ahead of print. PMID 41402044
- [Derived] Mathioudakis AG, Bate S, Sivapalan P, Jensen JS, Singh D, Vestbo J. Rethinking Blood Eosinophils for Assessing Inhaled Corticosteroids Response in COPD: A Post Hoc Analysis From the FLAME Trial. Chest. 2024 Nov;166(5):987-997. doi: 10.1016/j.chest.2024.06.3790. Epub 2024 Jul 9. PMID 38992490
- [Derived] Mackay AJ, Kostikas K, Roche N, Frent SM, Olsson P, Pfister P, Gupta P, Patalano F, Banerji D, Wedzicha JA. Impact of baseline symptoms and health status on COPD exacerbations in the FLAME study. Respir Res. 2020 Apr 22;21(1):93. doi: 10.1186/s12931-020-01354-8. PMID 32321518
- [Derived] Wedzicha JA, Singh D, Tsiligianni I, Jenkins C, Fucile S, Fogel R, Shen S, Goyal P, Mezzi K, Kostikas K. Treatment response to indacaterol/glycopyrronium versus salmeterol/fluticasone in exacerbating COPD patients by gender: a post-hoc analysis in the FLAME study. Respir Res. 2019 Jan 8;20(1):4. doi: 10.1186/s12931-019-0972-7. PMID 30621717
- [Derived] Frent SM, Chapman KR, Larbig M, Mackay A, Fogel R, Gutzwiller FS, Shen S, Patalano F, Banerji D, Kostikas K, Wedzicha JA. Capturing Exacerbations of Chronic Obstructive Pulmonary Disease with EXACT. A Subanalysis of FLAME. Am J Respir Crit Care Med. 2019 Jan 1;199(1):43-51. doi: 10.1164/rccm.201801-0038OC. PMID 30019939
- [Derived] Anzueto AR, Kostikas K, Mezzi K, Shen S, Larbig M, Patalano F, Fogel R, Banerji D, Wedzicha JA. Indacaterol/glycopyrronium versus salmeterol/fluticasone in the prevention of clinically important deterioration in COPD: results from the FLAME study. Respir Res. 2018 Jun 20;19(1):121. doi: 10.1186/s12931-018-0830-z. PMID 29925383
- [Derived] Roche N, Chapman KR, Vogelmeier CF, Herth FJF, Thach C, Fogel R, Olsson P, Patalano F, Banerji D, Wedzicha JA. Blood Eosinophils and Response to Maintenance Chronic Obstructive Pulmonary Disease Treatment. Data from the FLAME Trial. Am J Respir Crit Care Med. 2017 May 1;195(9):1189-1197. doi: 10.1164/rccm.201701-0193OC. PMID 28278391
- [Derived] Wedzicha JA, Banerji D, Chapman KR, Vestbo J, Roche N, Ayers RT, Thach C, Fogel R, Patalano F, Vogelmeier CF; FLAME Investigators. Indacaterol-Glycopyrronium versus Salmeterol-Fluticasone for COPD. N Engl J Med. 2016 Jun 9;374(23):2222-34. doi: 10.1056/NEJMoa1516385. Epub 2016 May 15. PMID 27181606

RESULTS

PARTICIPANT FLOW:
Groups:
- Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS): Salmeterol/fluticasone (50/500μg) twice a day
Period: Planned Treatment Epoch
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Started | 1680 | 1682
Full Analysis Set (FAS) | 1675 | 1679
Per-protocol Set (PPS) | 1528 | 1556
Serial Spirometry Set | 280 | 279
Safety Set (SAF) | 1678 | 1680
Urine Cortisol Set | 266 | 269
Completed | 1478 | 1474
Not Completed | 202 | 208
Not completed — Subject/guardian decision | 149 | 151
Not completed — Death | 29 | 30
Not completed — Physician Decision | 18 | 16
Not completed — Protocol deviation | 2 | 3
Not completed — Lost to Follow-up | 4 | 4
Not completed — Technical problems | 0 | 4
Period: Double-blind Treatment
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Started | 1678 | 1680
Completed | 1400 | 1360
Not Completed | 278 | 320
Not completed — Adverse Event | 129 | 145
Not completed — Subject/guardian decision | 111 | 125
Not completed — Lack of Efficacy | 17 | 22
Not completed — Physician Decision | 13 | 16
Not completed — Protocol deviation | 8 | 7
Not completed — Technical problems | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS) | Total
Number analyzed (Participants) | 1680 | 1682 | 3362
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (7.89) | 64.5 (7.70) | 64.6 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 381 | 424 | 805
  Male | 1299 | 1258 | 2557

OUTCOME MEASURES:

1. Primary Outcome: Rate of COPD Exacerbations
Description: COPD exacerbations starting between first dose and one day after last treatment are included. COPD exacerbations that occurred within 7 days of each other are collapsed as one event. Estimates are from a generalized linear model assuming a negative binomial distribution with terms for treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region. As the offset variable log(exposure time in years) was used.
Time Frame: 52 weeks
Population: The per-protocol set (PPS) included all patients in the FAS without any major protocol deviations. Only PPS patients with non-missing values for all terms in negative binomial model are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD Exacerbations/year
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1528 | 1556
COPD Exacerbations/year | 3.59 [3.28 to 3.94] | 4.03 [3.68 to 4.41]
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Non-Inferiority or Equivalence — Study was designed to have >95% power to rule out a 1.15-fold increase in the rate exacerbations for QVA149 vs. salmeterol/fluticasone; Generalized linear model; Rate Ratio = 0.89, 95% CI 2-sided [0.83 to 0.96] — If the upper limit of the confidence interval was <1.15 then non-inferiority of QVA149 compared to SFC could be claimed
Statistical Analysis 2: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p = 0.003, Generalized linear method; Rate Ratio = 0.89, 95% CI 2-sided [0.83 to 0.96] — If non-inferiority was demonstrated, superiority of QVA149A compared to SFC in reducing exacerbation rate could be claimed if the upper limit of the same CI was less than 1

2. Secondary Outcome: Time to First COPD Exacerbation.
Description: First COPD exacerbations starting between first dose and one day after last treatment are included. Cox regression model includes terms for treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region.
Time Frame: 52 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug and had no major GCP violations. Only FAS patients with non-missing values for all terms in Cox regression model are included.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Days | 71.0 [60.0 to 82.0] | 51.0 [46.0 to 57.0]
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.78 to 0.91]

3. Secondary Outcome: Rate of Moderate to Severe COPD Exacerbations.
Description: COPD exacerbations starting between date of first dose and one day after last treatment are included. COPD exacerbations that occurred within 7 days of each other are collapsed as one event with the worst severity. A COPD exacerbation of moderate severity meets the symptoms definition in the protocol and requires treatment with systemic corticosteroids and/or antibiotics. A severe COPD exacerbation requires hospitalization. Estimates are from a generalized linear model assuming a negative binomial distribution with terms for treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region. The offset variable log(exposure time in years) was used.
Time Frame: 52 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug and had no major GCP violations. Only FAS patients with non-missing values for all terms in negative binomial model are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD Exacerbation/year
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1651 | 1656
COPD Exacerbation/year | 0.98 [0.88 to 1.10] | 1.19 [1.07 to 1.32]
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p < 0.001, Generalized linear model; Rate Ratio = 0.83, 95% CI 2-sided [0.75 to 0.91]

4. Secondary Outcome: Time to First Moderate to Severe COPD Exacerbation.
Description: as for outcome 2
Time Frame: 52 weeks.
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug and had no major GCP violations. Only FAS patients with non-missing values for all terms in the Cox regression model are included.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Days | NA [NA to NA] — NA -Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated | 308.0 [283.0 to 352.0]
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.70 to 0.86]

5. Secondary Outcome: Rate of Moderate to Severe COPD Exacerbations Requiring Treatment With Systemic Corticosteroids
Description: COPD exacerbations starting between date of first dose and one day after last treatment are included. COPD exacerbations that occurred within 7 days of each other are collapsed as one event with the worst severity. Estimates are from a generalized linear model assuming a negative binomial distribution with fixed effects of treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region. The offset variable log(exposure time in years) was used.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD Exacerbation/year
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1651 | 1656
COPD Exacerbation/year | 0.18 [0.14 to 0.22] | 0.18 [0.14 to 0.23]

6. Secondary Outcome: Rate of Moderate to Severe COPD Exacerbations Requiring Treatment With Antibiotics
Description: Estimates are from a generalized linear model assuming a negative binomial distribution with terms for treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region. The offset variable log(exposure time in years) was used. COPD exacerbations starting between first dose and one day after last treatment are included .
Time Frame: 52 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug. Only FAS patients with non-missing values for all terms in negative binomial model are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD Exacerbation/year
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1651 | 1656
COPD Exacerbation/year | 0.17 [0.13 to 0.22] | 0.22 [0.17 to 0.28]

7. Secondary Outcome: Rate of Moderate to Severe COPD Exacerbations Requiring Hospitalization. COPD Exacerbations Starting Between First Dose and One Day After Last Treatment Are Included.
Description: All exacerbations requiring hospitalization are considered severe according to protocol definitions so this is the rate of severe COPD exacerbations only. Note - an ER visit of longer than 24 hours was considered a hospitalization.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD Exacerbation/year
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1651 | 1656
COPD Exacerbation/year | 0.15 [0.11 to 0.19] | 0.17 [0.13 to 0.22]

8. Secondary Outcome: Rate of Moderate to Severe COPD Exacerbations Requiring Re-hospitalization Within 30 Days
Description: Re-hospitalizations are defined as hospitalizations starting within the first 30 days after a severe COPD exacerbation and between first dose and one day after date of last treatment. Generalized linear model assuming a negative binomial distribution with terms for treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region. The offset variable log(exposure time in years) was used. COPD exacerbations starting between first dose and one day after last treatment are included.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: COPD Exacerbation/year
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
COPD Exacerbation/year | 0.0 (0.15) | 0.0 (0.12)

9. Secondary Outcome: Time to First Moderate to Severe COPD Exacerbations Requiring Treatment With Systemic Corticosteroids
Description: Cox regression model includes terms for treatment, baseline total symptom score, baseline COPD exacerbation history (i.e. number of COPD exacerbations during the past 12 months prior to study), smoking status at screening, ICS use at screening, airflow limitation severity, and region. COPD exacerbations starting between first dose and one day after date of last treatment are included.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Days | NA [NA to NA] — NA- Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated | NA [NA to NA] — NA- Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p = 0.256, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.74 to 1.08]

10. Secondary Outcome: Time to First Moderate to Severe COPD Exacerbations Requiring Treatment With Antibiotics
Description: as for outcome 9
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Days | NA [NA to NA] — NA- Parameters not estimated, data did not reach median | NA [NA to NA] — NA- Parameters not estimated, data did not reach median
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p = 0.008, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.69 to 0.95]

11. Secondary Outcome: Time to First Moderate to Severe COPD Exacerbations Requiring Hospitalization
Description: as for outcome 9
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Days | NA [NA to NA] — NA- Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated | NA [NA to NA] — NA- Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p = 0.046, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00]

12. Secondary Outcome: Time to First Moderate to Severe COPD Exacerbations Requiring Re-hospitalization Within 30 Days
Description: as for outcome 9
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Days | NA [NA to NA] — NA- Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated | NA [NA to NA] — NA- Parameters not estimated since less than 50% of the patients had an event, the median could not be calculated
Statistical Analysis 1: Comparison: QVA149 vs Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS); Test type: Superiority or Other; p = 0.790, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.38 to 2.10]

13. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: Change from baseline. Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, airflow limitation severity, region, visit, treatment-by-visit interaction, and baseline FEV1-by-visit interaction.
Time Frame: Baseline, day 1 (30 min and one hour post dose)
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug and did not have any major GCP violations. Only FAS patients with non-missing values for all terms in MMRM are included.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Liters
  Day 1, 30 min post-dose (n=1659, 1663) | 0.121 (0.0049) | 0.076 (0.0049)
  Day 1, one hour post-dose (n=1657, 1664) | 0.147 (0.0054) | 0.092 (0.0054)

14. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: Change from baseline in trough value. Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, airflow limitation severity, visit, treatment-by-visit interaction, and baseline FEV1-by-visit interaction.
Time Frame: Baseline, 4 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug and no major GCP violations. Only FAS patients with non-missing values for all terms in MMRM are included.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1597 | 1595
Liters | 0.079 (0.0070) | 0.006 (0.0070)

15. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: as for outcome 14
Time Frame: Baseline, 12 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug and had no major GCP violations. Only FAS patients with non-missing values for all terms in MMRM are included.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1597 | 1595
Liters | 0.070 (0.0072) | -0.008 (0.0072)

16. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: as for outcome 14
Time Frame: Baseline, 26 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1597 | 1595
Liters | 0.049 (0.0073) | -0.037 (0.0074)

17. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: as for outcome 14
Time Frame: Baseline, 38 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1597 | 1595
Liters | 0.034 (0.0074) | -0.039 (0.0075)

18. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: as for outcome 14
Time Frame: Baseline, 52 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1597 | 1595
Liters | 0.015 (0.0075) | -0.048 (0.0076)

19. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second AUC (0-12h)
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, baseline FEV1 * visit interaction, and visit, treatment * visit interaction. The trapezoidal rule was used to calculate FEV1 AUC and then normalized to the length of time"
Time Frame: Baseline, 52 weeks
Population: Serial spirometry set - Serial spirometry set includes the patients who performed additional serial spirometry, a subset of FAS. Only patients with non-missing values for all terms in MMRM are included.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 279 | 277
Liters | 0.078 (0.0174) | -0.032 (0.0176)

20. Secondary Outcome: Change From Baseline in Total St. George's Respiratory Questionnaire Score
Description: The St. George Respiratory Questionnaire C (SGRQ-C) is a disease-specific measure of health status for use in COPD that was used to provide the health status measurements in this study. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline SGRQ-C total score, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, airflow limitation severity, visit, treatment*visit Interaction, baseline SGRQ-C total score*visit + region. lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of health status. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug. Only FAS patients with non-missing values for all terms in MMRM are included.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1602 | 1593
Score on a scale | -2.3 (0.36) | -2.3 (0.36)

21. Secondary Outcome: Change From Baseline in Total St. George's Respiratory Questionnaire Score
Description: as for outcome 20
Time Frame: Baseline, 12 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1602 | 1593
Score on a scale | -3.2 (0.38) | -1.9 (0.38)

22. Secondary Outcome: Change From Baseline in Total St. George's Respiratory Questionnaire Score
Description: as for outcome 20
Time Frame: Baseline, 26 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1602 | 1593
Score on a scale | -3.5 (0.39) | -2.3 (0.39)

23. Secondary Outcome: Change From Baseline in Total St. George's Respiratory Questionnaire Score
Description: as for outcome 20
Time Frame: Baseline, 38 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1602 | 1593
Score on a scale | -3.5 (0.40) | -1.7 (0.40)

24. Secondary Outcome: Change From Baseline in Total St. George's Respiratory Questionnaire Score
Description: as for outcome 20
Time Frame: Baseline, 52 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1602 | 1593
Score on a scale | -3.1 (0.41) | -1.9 (0.41)

25. Secondary Outcome: Change From Baseline in the Number of Puffs of Rescue Medication
Description: A linear mixed model (LMM) was used for this analysis Change from baseline in mean number of puffs. LMM including: treatment, baseline value, smoking status at screening, ICS use at screening, airflow limitation severity, region and random effect of center nested within region.
Time Frame: Baseline, 52 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug. Only FAS patients with non-missing values for all terms in LLM are included.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs per day
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1675 | 1679
Number of puffs per day | -1.01 (0.097) | -0.76 (0.097)

26. Secondary Outcome: Change From Baseline in the Safety of QVA149 ((110/50 μg o.d.) vs Fluticasone/Salmeterol (500/50μg Bid) in Terms of HPA Axis Function, as Determined by Collection of 24-hour Urine Cortisol.
Description: Urine cortisol/creatinine ratio
Time Frame: Baseline, 52 Weeks
Population: Urine cortisol set is the subset of patients who were measured with 24-hour Urine cortisol, a subset of safety set. The safety set included all patients who received at least one dose of study drug. At the post-baseline timepoint only patients with a value at both baseline and the post-baseline timepoint are included.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 162 | 154
ng/mL | 5.615 (26.633) [-96.93 to 509.17] | -10.390 (54.428) [-97.76 to 4444.65]

27. Secondary Outcome: Change From Baseline in Forced Vital Capacity
Description: Change from baseline in trough value (average of values measured 45 and 15 minutes prior to the morning dose). Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FVC was defined as the average of the pre-dose FVC measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FVC measurements, smoking status at screening, screening inhaled corticosteroid (ICS) use, region, baseline FVC * visit interaction, and visit, treatment * visit interaction
Time Frame: 4 Weeks, 12 Weeks, 26 Weeks, 38 Weeks, 52 Weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1597 | 1595
Liters
  4 weeks | 0.146 (0.0127) | -0.032 (0.0128)
  12 weeks | 0.134 (0.0131) | -0.071 (0.0131)
  26 weeks | 0.088 (0.0135) | -0.121 (0.0136)
  38 weeks | 0.071 (0.0137) | -0.111 (0.0137)
  52 weeks | 0.022 (0.0139) | -0.138 (0.0140)

28. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events, and Death
Description: The overall rate of adverse events reported from initiation through 30 days post last dose.
Time Frame: 52 weeks of treatment + 30 days
Population: The Safety set:all patients that received at least one dose of study medication and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received. The statement that a patient had no AEs also constituted a safety assessment. Only deaths occurring on treatment + 30 days after end of treatment were included
Measure: Number; unit: Number of participants
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Number analyzed (Participants) | 1678 | 1680
Number of participants
  Patients with at least one SAEs | 308 | 334
  Patients with at least one AE | 1459 | 1498
  Death | 24 | 24

ADVERSE EVENTS:
Arm/Group | QVA149 | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS)
Serious Adverse Events (participants affected / at risk) | 308/1678 | 334/1680
Other Adverse Events (participants affected / at risk) | 1363/1678 | 1424/1680
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=1678) | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS) (N=1680)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 2
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 4 | 2
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 1 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 5 | 7
ATRIAL FLUTTER (Cardiac disorders) | 2 | 3
ATRIAL TACHYCARDIA (Cardiac disorders) | 2 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 5 | 1
CARDIAC FAILURE (Cardiac disorders) | 5 | 7
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 3
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 3
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
COR PULMONALE (Cardiac disorders) | 0 | 2
COR PULMONALE CHRONIC (Cardiac disorders) | 0 | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 2
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 6 | 5
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 2
MYOCARDIAL RUPTURE (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 | 0
PROGRESSIVE CEREBELLAR DEGENERATION (Congenital, familial and genetic disorders) | 1 | 0
GOITRE (Endocrine disorders) | 1 | 1
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 | 1
OPHTHALMOPLEGIA (Eye disorders) | 1 | 0
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 1 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
ACID PEPTIC DISEASE (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
FAECALOMA (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 3
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 | 4
NAUSEA (Gastrointestinal disorders) | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 2 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 3
STOMATITIS (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
LOCAL SWELLING (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 1 | 1
PYREXIA (General disorders) | 1 | 2
SUDDEN CARDIAC DEATH (General disorders) | 1 | 1
SUDDEN DEATH (General disorders) | 1 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 2 | 0
HEPATIC CYST RUPTURED (Hepatobiliary disorders) | 0 | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0
FOOD ALLERGY (Immune system disorders) | 1 | 0
ABSCESS JAW (Infections and infestations) | 1 | 0
ABSCESS LIMB (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 1
ATYPICAL MYCOBACTERIAL INFECTION (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 4
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 2 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 1
ECZEMA INFECTED (Infections and infestations) | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 2
GASTROENTERITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 1 | 0
H1N1 INFLUENZA (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 1
INFECTED SKIN ULCER (Infections and infestations) | 1 | 0
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 2 | 0
INFECTIVE ANEURYSM (Infections and infestations) | 1 | 0
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 1
INFLUENZA (Infections and infestations) | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 7
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 3
MENINGITIS VIRAL (Infections and infestations) | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 2
ORAL VIRAL INFECTION (Infections and infestations) | 1 | 0
OTITIS EXTERNA (Infections and infestations) | 1 | 0
OTITIS MEDIA CHRONIC (Infections and infestations) | 1 | 0
PERITONITIS (Infections and infestations) | 1 | 2
PHARYNGITIS (Infections and infestations) | 1 | 0
PNEUMOCOCCAL INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 34 | 54
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 1
PSEUDOMONAS INFECTION (Infections and infestations) | 0 | 1
PULMONARY SEPSIS (Infections and infestations) | 4 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 1
SINUSITIS (Infections and infestations) | 2 | 1
SPUTUM PURULENT (Infections and infestations) | 0 | 1
TUBERCULOUS PLEURISY (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 9 | 15
URETERITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 1 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 0 | 1
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 | 2
OVERDOSE (Injury, poisoning and procedural complications) | 2 | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
WOUND DECOMPOSITION (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2
BLOOD POTASSIUM INCREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 1
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 3
DIET REFUSAL (Metabolism and nutrition disorders) | 1 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 2 | 0
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
ADRENAL GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HYPOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LARGE INTESTINE BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
MALIGNANT MESENCHYMOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PENILE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
URETHRAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL GANGLIA STROKE (Nervous system disorders) | 0 | 1
BRAIN INJURY (Nervous system disorders) | 1 | 0
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 0 | 1
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 | 0
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 | 1
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 0 | 1
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
CEREBRAL THROMBOSIS (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 2
CLUSTER HEADACHE (Nervous system disorders) | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 1
EPILEPSY (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 2 | 0
LACUNAR INFARCTION (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 2 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 1
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1
DELIRIUM TREMENS (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
HALLUCINATION (Psychiatric disorders) | 1 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 2 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 2
TESTICULAR TORSION (Reproductive system and breast disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 5 | 4
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOPLEURAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 182 | 207
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 4
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 5
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 2
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HILAR ENLARGEMENT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 11 | 6
LINEAR IGA DISEASE (Skin and subcutaneous tissue disorders) | 0 | 1
PARAPSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 2 | 3
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 | 1
AORTIC CALCIFICATION (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 0
EMBOLISM ARTERIAL (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 3 | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0
LERICHE SYNDROME (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 4 | 0
PERIPHERAL EMBOLISM (Vascular disorders) | 0 | 1
TEMPORAL ARTERITIS (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 1
VARICOSE ULCERATION (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=1678) | Long Acting B2 Agonist (LABA) and Inhaled Corticosteroid (ICS) (N=1680)
CONSTIPATION (Gastrointestinal disorders) | 19 | 17
DIARRHOEA (Gastrointestinal disorders) | 19 | 24
DYSPEPSIA (Gastrointestinal disorders) | 18 | 9
GASTRITIS (Gastrointestinal disorders) | 10 | 20
NON-CARDIAC CHEST PAIN (General disorders) | 20 | 11
OEDEMA PERIPHERAL (General disorders) | 26 | 13
PYREXIA (General disorders) | 17 | 27
BRONCHITIS (Infections and infestations) | 29 | 41
GASTROENTERITIS (Infections and infestations) | 10 | 18
INFLUENZA (Infections and infestations) | 34 | 55
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 76 | 91
NASOPHARYNGITIS (Infections and infestations) | 197 | 194
ORAL CANDIDIASIS (Infections and infestations) | 20 | 71
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 2 | 17
PNEUMONIA (Infections and infestations) | 19 | 27
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 17 | 8
RHINITIS (Infections and infestations) | 27 | 28
SINUSITIS (Infections and infestations) | 16 | 20
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 79 | 82
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 121 | 157
URINARY TRACT INFECTION (Infections and infestations) | 14 | 22
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 131 | 136
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 20 | 23
BACK PAIN (Musculoskeletal and connective tissue disorders) | 35 | 34
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 17 | 13
DIZZINESS (Nervous system disorders) | 6 | 27
HEADACHE (Nervous system disorders) | 38 | 34
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1262 | 1331
COUGH (Respiratory, thoracic and mediastinal disorders) | 50 | 49
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 7 | 30
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 41 | 47
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 35 | 33
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 10 | 23
HYPERTENSION (Vascular disorders) | 44 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.